CLINICAL TRIAL: NCT05251753
Title: Evaluation of a Novel Sutureless Drain Securement Device (K-Lock Device) and Comparison to Standard Suture-based Drain Securement Techniques
Brief Title: Evaluation of a Novel Sutureless Drain Securement Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00080041
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-01

CONDITIONS: Skin Injury
Keywords: drain; suture; body contouring

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- A K-Lock left (Experimental): A) left side K-Lock with right side suture-based technique
  Interventions: Device: K-Lock
- B K-Lock right (Experimental): B) right side K-Lock with left side suture-based technique.
  Interventions: Device: K-Lock

INTERVENTIONS:
Device: K-Lock — Patients will be randomized to either A) left side K-Lock with right side suture-based technique or B) right side K-Lock with left side suture-based technique.

SUMMARY:
The purpose of this study is to evaluate an investigational sutureless drain securement device (K-Lock) and compare this device to standard drain securement.

DETAILED DESCRIPTION:
This study will evaluate the feasibility, safety and efficacy of a novel sutureless drain securement device (K-Lock) via direct comparison to suture-based techniques. In this study the sutureless drain securement device will be compared to the use of sutures to secure drains. Patients will be randomized to either A) left side K-Lock with right side suture-based technique or B) right side K-Lock with left side suture-based technique.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Patient of the Department of Plastic and Reconstructive Surgery
* Able to sign English language Consent form
* Undergoing any of the following procedures requiring placement of 2 or more drains (preferably bilateral) including: Breast reconstruction, Bilateral Breast Reduction, Abdominoplasty, Body Contour surgery (e.g. panniculectomy, brachiplasty, thighplasty)

Exclusion Criteria:

* Patients with unilateral drain placement
* Unable to sign English language consent form
* Allergy to Tegaderm Dressing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2025-03-06 (Actual); Study Completion 2025-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa David, MD MBA, Principal Investigator — Wake Forest University Health Sciences; Adam J Katz, MD, Study Director — Wake Forest University Health Sciences
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A K-Lock Left | B K-Lock Right
Started | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A K-Lock Left | B K-Lock Right | Total
Number analyzed (Participants) | 13 | 9 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.30769231 (8.606050346) | 42.77777778 (15.03144851) | 44.27272727 (11.40251358)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 9 | 22

OUTCOME MEASURES:

1. Primary Outcome: Time it Takes to Secure and Dress Each Drain in Totality
Description: Time it takes to secure and dress each drain will be evaluated in totality by evaluation of video recordings to record timestamps and documented on "K-Lock Study Outcomes" tool. This will help determine the feasibility of using this device.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | A K-Lock Left | B K-Lock Right
Number analyzed (Participants) | 13 | 9
Seconds
  Time to secure K-Lock and dress | 67 (0.013750872) | 79 (0.031915706)
  Time to secure Suture and dress | 114 (0.018172119) | 94 (0.012821128)

2. Secondary Outcome: Ease of Use
Description: For each participant, the surgeon will evaluate the K-Lock device ease of use of on a scale from 1-5. A higher score indicates greater ease of use.
Time Frame: Day of Surgery
Population: Surgeons were assessed for this Outcome Measure but were not enrolled in the study. It was pre-specified to collect and report the scores for the K-Lock device itself, regardless of left or right. Individual surgeons performed surgery on more than one participant which explains why the number of surgeries is higher than the number of surgeons (overall number of participants analyzed).
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: surgeries
Groups:
- Surgeons: Surgeons that assessed of use for K-Lock device
Arm/Group | Surgeons
Number analyzed (Participants) | 6
Number analyzed (surgeries) | 13
score on a scale | 4.553846154 (0.224256939)

3. Secondary Outcome: Skin Injury
Description: Skin Injury will be evaluated by inspecting device sites for instances of skin injury at each office visit and will be recorded on "K-Lock Study Outcomes" tool. Skin Injury will also be evaluated by quantitative feedback obtained in the "Drain Securement Survey" given to patients post-operatively. Number of Injuries for all K-Lock sites will be reported as a total.
Time Frame: On Average Day 10
Measure: Number; unit: Occurrence of skin injury
Units Other Than Participants: K-Lock Drain Sites
Groups:
- K-Lock Drain Sites: Every K-Lock Drain Site
Arm/Group | K-Lock Drain Sites
Number analyzed (Participants) | 22
Number analyzed (K-Lock Drain Sites) | 22
Occurrence of skin injury | 1

ADVERSE EVENTS:
Time Frame: 3 months
Description: Reported all Adverse Events within 24 hours of becoming aware.
Arm/Group | A K-Lock Left | B K-Lock Right
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/9
Other Adverse Events (participants affected / at risk) | 1/13 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A K-Lock Left (N=13) | B K-Lock Right (N=9)
Device became loose (Surgical and medical procedures) | 1 (1) | 0 (0) — Patient called the triage nurse to report that the device had become loose. Patient was brought in to be examined and device was removed. Drain was secured with suture.
Hematoma (Surgical and medical procedures) | 0 (0) | 1 (1) — Patient taken back to OR for evaluation of a hematoma and the device was removed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/53/NCT05251753/Prot_SAP_000.pdf
  • Informed Consent Form (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT05251753/ICF_001.pdf